CLINICAL TRIAL: NCT03216317
Title: Effect of Handgrip's Isometric Training on Blood Pressure and on the Autonomic Modulation of Hypertense Individuals at the Basic Health Units: A Multicentric Study
Brief Title: Isometric Training on Blood Pressure and on the Autonomic Modulation of Hypertensive Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Israelita Albert Einstein (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 55555
Record Dates: First submitted 2017-07-11; First posted 2017-07-13 (Actual); Last update posted 2019-02-08 (Actual); Status verified 2017-07

CONDITIONS: Hypertension
Keywords: Hypertension; Hypotension; Cardiovascular system
MeSH Terms: conditions — Hypertension; Hypotension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Active Comparator): Subjects will perform three weekly sessions of isometric handgrip training consisting of four series (two in each arm) with two minutes of isometric contraction with intensity of 30% of maximum voluntary contraction with interval between the two-minute series under the guidance of the trained researcher.
  Interventions: Behavioral: Intervention Group
- Control Group (No Intervention): Individuals randomized to Control Group will be encouraged to increase their level of general physical activity, but without specific recommendations on physical activity.

INTERVENTIONS:
Behavioral: Intervention Group — Isometric handgrip training consisting of four series
  Arms: Intervention Group

SUMMARY:
Objective: analyze the effects of isometric handgrip exercise on arterial pressure and on the autonomic cardiac modulation of hypertensive individuals treated in the Unified Health System (UHS).

Intervention: Patients were randomized into Supervised group (SG) and control group (CG). SG will perform supervised isometric handgrip exercise for three weekly sessions in four sets with two minutes of isometric contraction with 30% of maximal voluntary contraction (MVC), In CG, individuals will be encouraged to increase their level of physical activity.

Measurements: Blood pressure, autonomic modulation

DETAILED DESCRIPTION:
The objective of this study is to analyze the effects of isometric handgrip exercise on arterial pressure and on the autonomic cardiac modulation of hypertensive individuals treated in the Unified Health System (UHS). Two prospective, randomized, controlled trials will be conducted with hypertensive patients in the public health network of Petrolina (PE) and São Paulo (SP). Included in the study will be individuals with an age group over 18 years of both genders, with systemic arterial hypertension (SAH) controlled with the use of antihypertensive medication, non-smokers and without the presence of diabetes or other cardiovascular diseases that will be allocated randomly in two groups: supervised group (SG) and control group (CG). SG will be instructed to perform supervised isometric handgrip exercise for three weekly sessions in four sets with two minutes of isometric contraction with 30% of maximal voluntary contraction (MVC) of the subjects and interval between two-minute series. In CG, individuals will be encouraged to increase their level of physical activity. Prior to initiation and after 12 weeks of intervention, blood pressure, autonomic cardiac modulation and level of physical activity will be obtained.

ELIGIBILITY:
Inclusion Criteria:

* It will include individuals with age range over 18 years of both genders and with controlled hypertension using antihypertensive medication and without the presence of diabetes or other cardiovascular diseases and who do not present high cardiovascular risk.

Exclusion Criteria:

* Those individuals who: a) are diagnosed of diseases such as dyslipidemia, diabetes mellitus, cardiovascular or pulmonary diseases; B) adhere to another program of physical activities besides the training offered by the present study; C) change the class and dose of medication during the study; and d) aggravate the disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2017-07-15 (Actual); Primary Completion 2017-12-30 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
Blood Pressure measure | 12 weeks
  The subjects will remain for ten minutes in the seated position, following the guidelines of the VII Brazilian Direction of Hypertension. Three consecutive measurements, one minute apart, in the non-dominant arm and with a cuff size suitable for the circumference of the arm will be performed. The value used will be the average of the last two measures, as recommended by the VII Brazilian Arterial Hypertension Guideline.

SECONDARY OUTCOMES:
Heart rate variability measure | 12 weeks
  The patients will remain 10 minutes lying down, during which the heart rate variability (HRV) intervals will be registered, using a valid heart rate monitor for this function (RS800CX, Polar Electro, Finland). It will be considered a valid signal those with at least five minutes of signal stationary.

CONTACTS AND LOCATIONS:
Overall Officials: Raphael MR Dias, PhD, Principal Investigator — Hospital Israelita Albert Einstein
Locations (1):
- Unidade Básica de Saúde, Petrolina, Pernambuco, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carlson DJ, Dieberg G, Hess NC, Millar PJ, Smart NA. Isometric exercise training for blood pressure management: a systematic review and meta-analysis. Mayo Clin Proc. 2014 Mar;89(3):327-34. doi: 10.1016/j.mayocp.2013.10.030. PMID 24582191
- [Background] Inder JD, Carlson DJ, Dieberg G, McFarlane JR, Hess NC, Smart NA. Isometric exercise training for blood pressure management: a systematic review and meta-analysis to optimize benefit. Hypertens Res. 2016 Feb;39(2):88-94. doi: 10.1038/hr.2015.111. Epub 2015 Oct 15. PMID 26467494
- [Derived] Palmeira AC, Farah BQ, Silva GOD, Moreira SR, Barros MVG, Correia MA, Cucato GG, Ritti-Dias RM. Effects of isometric handgrip training on blood pressure among hypertensive patients seen within public primary healthcare: a randomized controlled trial. Sao Paulo Med J. 2021 Nov 15;139(6):648-656. doi: 10.1590/1516-3180.2020.0796.R1.22042021. eCollection 2021. PMID 34787298